CLINICAL TRIAL: NCT04285450
Title: The Clinical Effect of Vitamin K Administration in Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amani Mohamed, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL2182
Record Dates: First submitted 2019-10-17; First posted 2020-02-26 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vitamin K

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin K 1mg (Experimental)
  Interventions: Dietary Supplement: Vitamin K
- Control (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin K — 1mg
  Arms: Vitamin K 1mg
Other: Placebo — Lactose
  Arms: Control

SUMMARY:
The aim of this study is to examine the possible clinical effects associated with vitamin K supplementation on the glycemic control, insulin sensitivity and lipid profile of type II diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 21-65 years old diagnosed with Type II diabetes.
* Fasting blood glucose concentration ≥ 126 mg/dL .
* Normal liver Function tests defined as ALT levels up to 33 U/L for males and up to 25 U/L for females, Albumin levels ≥ 3.5 g/dL, Bilirubin up to 1.1 mg/dL .
* Normal clotting function defined as defined by INR.
* Normal kidney function defined as serum creatinine values up to 1.3 mg/dL.

Exclusion Criteria:

* Type I diabetic patients.
* Use of supplements with potential effect on vitamin K level namely supplements containing vitamin K, co-enzyme Q10 or vitamin E > 400 IU .
* Patients requiring anti-coagulant therapy including patients with prosthetic valves, mitral tissues, DVT, PE, atrial fibrillation and valvular heart disease.
* Patient with history of coagulation, MI, stroke and embolization.
* Pregnant or breast feeding women.
* Being on hormonal therapy or receiving contraceptive pills.
* Patients treated with glucocorticoids, thiazide diuretics, and atypical antipsychotics.
* Patients on cholestyramine, antibiotics and coumarins.
* Patients on lipid lowering agents.
* Known intestinal malabsorption syndrome, cholestasis or steatorrhea.
* Smokers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2019-10-27 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Homeostasis model assessment of insulin resistance (HOMA-IR) | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al Aini Hospital, Cairo, Egypt

REFERENCES:
- [Derived] Ali AM, Abbassi MM, Sabry NA, Fawzi M, Mousa S. The effect of vitamin K4 supplementation on insulin resistance in individuals with type 2 diabetes: a double-blind randomised placebo-controlled clinical trial. Eur J Nutr. 2023 Dec;62(8):3241-3249. doi: 10.1007/s00394-023-03215-8. Epub 2023 Aug 8. PMID 37552330